CLINICAL TRIAL: NCT04359511
Title: Efficacy and Safety of Corticosteroids in Oxygen-dependent Patients With COVID-19 Pneumonia in Grand Ouest Interregion France
Brief Title: Efficacy and Safety of Corticosteroids in Oxygen-dependent Patients With COVID-19 Pneumonia
Acronym: CORTICOVIDHUGO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: COMPETITOR TEST (RECOVERY)
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CORTI-COVID-19-HUGO; DR200136 (Registry Identifier: Sponsor ID)
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Prednisone; Hydrocortisone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- corticosteroid + Optimized Standard of Care (Experimental): * prednisone 0.7 mg/kg/day for 10 days, administered orally, once a day, or
  * hydrocortisone hemisuccinate 3.5 mg/kg/day by continuous infusion for 10 days, administered by IV route if the patient cannot take drugs by oral route,
    * standard of care
  Interventions: Drug: Prednisone; Drug: Hydrocortisone
- Optimized Standard of Care (No Intervention): standard of care

INTERVENTIONS:
Drug: Prednisone — prednisone 0.7 mg/kg/d (PO)
  Arms: corticosteroid + Optimized Standard of Care
Drug: Hydrocortisone — hémisuccinate d'hydrocortisone 3,5 mg/kg/jour (IV)
  Arms: corticosteroid + Optimized Standard of Care

SUMMARY:
To date, there is no efficient therapeutics to prevent or treat COVID-19 related pulmonary failure. Corticosteroids (CS) could be a helpful therapeutic. Retrospective reports suggested survival improvement in patients with acute respiratory distress syndrome (ARDS). CT scan for COVID19 hospitalized patients showed sometimes unusual aspects of pneumonia, suggestive of an organizing phase of diffuse alveolar damage (DAD).

We hypothesize that, in the context of alveolar aggression induced by COVID-19, CT scan could help to individualize patients with a high probability of pulmonary organizing process who could benefit from CS treatment.

DETAILED DESCRIPTION:
"Severe acute respiratory syndrome" coronavirus 2 (SARS-Cov-2) is a new coronavirus that induces pneumonia called Corona Virus Disease- 19 (COVID-19), an infected 1.5 million people worldwide and caused the more than 85,000 patients died. COVID-19 usually comes in the form of viral pneumonia but with the peculiarities of a risk frequent worsening towards acute respiratory distress syndrome (ARDS) and a usual duration of oxygen dependence in fragile patients by their age or their comorbidities. To date, there is no therapy effective in preventing or treating COVID-19. Drug identification is a major concern and a public health emergency. Retrospective study (Wu 2020) highlighted improved survival in COVID-19 patients with acute ARDS and treated with corticosteroids (CS). So even in the absence of evidence of effectiveness, the SCs are used for COVID-19 oxygen-dependent patients or with an ARDS. However, their benefit / risk remains debated (Russel 2020). On histological samples of COVID-19, diffuse alveolar damage (DAD) has been especially observed (Hanley 2020). DAD is described histologically in an exudative phase, an organizational phase and a irreversible fibrotic phase (Hughes 2017). SC could have an effect beneficial by limiting the exudative / inflammatory phase but also that organization whose histological and CT aspects are sometimes indistinguishable from organized pneumonia, a form of pulmonary repair aberrant very corticosensitive (Travis 2013). Chest scans performed in the face of the persistence or worsening of oxygen dependence beyond the 7th day of COVID-19 symptoms, could help discern indirect complications (pulmonary embolism, exacerbation of COPD, bacterial superinfection, etc.) of an unfavorable course COVID-19 (by displaying an aspect suggesting DAD in particular during the organization phase). We hypothesize that, in the context of COVID-19, the SCs may be beneficial in patients with CT scans thoracic images suggestive of DAD either at the exudative phase or at the pulmonary organization phase.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old,
* Hospitalized with a proven diagnosis of COVID-19 (SARS-CoV-2 positive in RTPCR), in medicine or in intensive care.
* With a need for oxygen therapy ≥ 2 l / min to maintain a Sp02> 92% or a need for oxygen therapy to maintain a PaO2 / FiO2> 300 mmHg (for intubated patients).
* With a chest scanner at least 7 days after the onset of symptoms, and whose centralized interpretation shows a CT scan aspect suggestive of intense and predominant DAD which can explain the patient's oxygen dependence.
* Signature of a free, written and informed consent by the patient, or the person of trust
* Affiliate or beneficiary of a social security scheme.

Exclusion Criteria:

* Patients already treated by CS for a chronic disease.
* Patients with a known contraindication to SC, such as hypersensitivity.
* Patients at risk of dying within 48 hours.
* Pregnant or breastfeeding women.
* Patients under guardianship, curatorship, safeguard of justice.
* Poor understanding of the French language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement defined by the improvement of 2 points on a 7-category ordinal scale, at 14 days. | 14 days
  The 7-category ordinal scale is as follow:
  1. Not hospitalized with resumption of usual activities
  2. Not hospitalized, but unable to resume usual activities
  3. Hospitalized, not requiring O2
  4. Hospitalized, requiring O2 from 1 to 5 l/min
  5. Hospitalized, requiring O2 >6 l/min, nasal high-flow O2, non-invasive mechanical ventilation, or both
  6. Hospitalized, requiring ECMO, invasive mechanical ventilation, or both
  7. Death.

SECONDARY OUTCOMES:
Proportion of patients free of oxygen at day 14 and 28 | 14 and 28 days
Proportion of patients discharged alive from hospital at day 14 and 28 | 14 and 28 days
Time to discharge for patients alive | 28 days
Proportion of patients that were hospitalized to ICU or who died at day 14 and 28 | 14 and 28 days
14 and 28 day mortality rate | 14 and 28 days
The time until weaning from oxygen therapy | 28 days
The proportion of patients with clinical degradation of at least 1 point on the ordinal scale to 7 categories on D14 and D28 | 14 and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: LOUIS BERNARD, MD, PhD, Principal Investigator — CHRU DE TOURS; JOUNEAU STEPHANE, MD, PhD, Principal Investigator — Rennes University Hospital; MAILLOT FRANCOIS, MD, Principal Investigator — CHRU DE TOURS; LIOGER BERTRAND, MD, Principal Investigator — CH DE BLOIS; GOUPIL FRANCOIS, MD, Principal Investigator — CH Le Mans; RABUT Thi- Tuyet Hong, MD, Principal Investigator — CH DE CHARTRES; POPA Mihai, MD, Principal Investigator — CH DE RDREUX; MOREL HUGUES, MD, Principal Investigator — CHR ORLEANS; GUY TIPHAINE, MD, Principal Investigator — CH DE VANNES; LEMMENS BRUNO, MD, Principal Investigator — CH AMBOISE; BAZIN YANN, MD, Principal Investigator — CH SAINT MALO; ROY XAVIER, MD, Principal Investigator — CH DE CHATEAUROUX; PECQUERIAUX OLIVIER, MD, Principal Investigator — CH DE BOURGES; MARCHAND ADAM Sylvain, MD, PhD, Principal Investigator — CHRU DE TOURS

IPD SHARING:
Plan to Share IPD: Undecided